CLINICAL TRIAL: NCT02201797
Title: Reproducibility and Repeatability of Multifunctional MRI Biomarkers of the Body
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Asan Medical Center (Other)
Collaborators: Bracco Diagnostics, Inc (Industry)
Responsible Party: Principal Investigator, Kyung Won Kim, Assistance Professor, Asan Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2014-0060
Record Dates: First submitted 2014-07-24; First posted 2014-07-28 (Estimated); Last update posted 2015-06-24 (Estimated); Status verified 2015-06

CONDITIONS: Metastatic Liver Cancer
Keywords: Reproducibility of Results; Liver neoplasm; Neoplasm metastasis; Regional Perfusion; Perfusion Magnetic Resonance Imaging
MeSH Terms: conditions — Liver Neoplasms; Neoplasm Metastasis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- DCE and DWI MRI (Experimental): MRI SCAN 1 and MRI SCAN 2 must be completed no less than 2 calendar days (to ensure 24 hours for clearance of gadolinium) and no greater than 14 days apart, and both must be completed prior to new treatment initiation. The same MRI unit and configuration must be used for MRI SCAN 1 and MRI SCAN 2.
  Interventions: Other: DCE MRI

INTERVENTIONS:
Other: DCE MRI

SUMMARY:
Advanced MRI (Magnetic Resonance Imaging) technique called DCE (Dynamic Contrast Enhanced) and DWI MRI can provide valuable information regarding tumor biology and response to treatment through various parameters. Validating stability of these parameters will further establish robustness and reliability of these promising biomarkers.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of metastatic liver cancer proven by pathology
* At least one liver tumor should be > 2cm in long diameter
* Patients with viable tumor proven in the other imaging modalities

Exclusion Criteria:

* Severe claustrophobia
* Presence of MRI-incompatible metallic objects or implanted medical devices in body
* Renal failure, as determined by glomerular filtration rate (GFR) < 30 mL/min/1.73 m2
* Weight greater than that allowable by the MRI table
* Chemotherapy within 28 days prior to enrollment
* Prior external radiation therapy to the liver, prior transarterial chemoembolization

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2014-10; Primary Completion 2015-06 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
repeatability coefficient (RC) | one year
  Repeatability coefficient of Ktrans, Kep, Ve, IAUGC60, and ADC value of the index tumor will be measured.

CONTACTS AND LOCATIONS:
Overall Officials: Kyung Won Kim, M.D., Principal Investigator — Asan Medical Center
Locations (1):
- Asan Medical Center, Seoul, South Korea